CLINICAL TRIAL: NCT04621409
Title: Effects of LEAP-2 on Postprandial Glucose Metabolism and Food Intake
Brief Title: LEAP2 on Postprandial Glucose Metabolism and Food Intake
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, head of department, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LEAP2
Record Dates: First submitted 2020-10-12; First posted 2020-11-09 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The study is designed as a clinical, placebo-controlled, double-blinded cross-over study involving two experimental study days.
Who Masked: Participant, Investigator
Masking Description: Day A and B will be conducted in a randomised, double-blinded order (blinded for the participant and the investigator) and noted by a third person not participating in the collection or analyses of data. The infusion order will be opened after the primary data analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- liver-enriched antimicrobial peptide 2 (Experimental): IV infusion of LEAP2, approximately 5 hours
  Interventions: Biological: Liver-enriched antimicrobial peptide 2
- Placebo (Placebo Comparator): IV infusion of saline, approximately 5 hours
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Liver-enriched antimicrobial peptide 2 — IV infusion of LEAP2, approximately 5 hours
  Arms: liver-enriched antimicrobial peptide 2
Biological: Placebo — IV infusion of saline, approximately 5 hours
  Arms: Placebo

SUMMARY:
The study aim to delineate the effects of the naturally occurring peptide liver-enriched antimicrobial peptide 2 (LEAP-2) on postprandial glucose metabolism and food intake in healthy volunteers. The overall objective is to investigate the physiological importance of LEAP-2 in healthy subjects.

DETAILED DESCRIPTION:
In a recent study, the molecular phenotype of enteroendocrine cells in the small intestine before and after Roux-en-Y Gastric Bypass (RYGB) surgery in obese individuals was examined. Enteroendocrine cells were identified and isolated from intestinal biopsies and analysed for differentially expressed genes by Illumina High Throughput RNA-sequencing. It was discovered that the gene encoding liver-enriched antimicrobial peptide 2 (LEAP-2), a naturally occurring peptide in humans, was significantly upregulated compared to baseline expression. Interestingly, LEAP-2 was recently shown to antagonize ghrelin function in response to feeding in mice. Moreover, the mature murine LEAP-2 peptide is identical in mice and humans. Thus, LEAP-2 has been identified as an endogenous peptide that may be able to alter feeding behaviour and maintenance of glucose levels during calorie restriction.

The study hypothesis is that LEAP-2 alters postprandial glucose metabolism and decreases appetite as well as food intake in relation to a liquid mixed meal and a standardised ad libitum meal compared with saline (placebo) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men
* Age between 18 and 25 years
* Body mass index between 20-35 kg/m2
* Informed consent

Exclusion Criteria:

* Anaemia (haemoglobin below normal range)
* Alanine aminotransferase (ALAT) and/or aspartate aminotransferase (ASAT) >2 times normal values) or history of hepatobiliary and/or gastrointestinal disorder(s)
* Nephropathy (serum creatinine above normal range and/or albuminuria)
* Allergy or intolerance to ingredients included in the standardised meals
* First-degree relatives with diabetes and/or glycated haemoglobin (HbA1c) >48 mmol/mol
* Regular tobacco smoking or use of other nicotine-containing products
* Any ongoing medication that the investigator evaluates would interfere with trial participation.
* Any physical or psychological condition that the investigator evaluates would interfere with trial participation including any acute or chronic illnesses

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Food intake | 260 to 290 minutes
  Difference in food intake during an ad libitum meal. Food intake is examined as kilojoules (kJ) and kJ/kg body weight of food eaten during the ad libitum meal.

SECONDARY OUTCOMES:
VAS | -30 to 290 minutes
  Visual analogue scales (VASs) assessing appetite, satiety and hunger sensations (from 0 to 10 cm on a scale = from mimimum to maximum sensation)
Alterations in gastric emptying | -30 to 290 minutes
  Paracetamol concentration in plasma after intake of 1.5 g paracetamol
Plasma insulin levels and beta cell secretion assessed by plasma C-peptide concentration relative to plasma glucose concentration | -30 to 290 minutes
  Plasma insulin levels and beta cell secretion assessed by plasma C-peptide concentration relative to plasma glucose concentration
Plasma/serum concentrations of LEAP-2, acyl-ghrelin as well as other glucose- and appetite-regulating gut hormones | -30 to 290 minutes
  Plasma/serum concentrations of LEAP-2, acyl-ghrelin as well as other glucose- and appetite-regulating gut hormones
Changes in resting energy expenditure (REE) | -30 to 290 minutes
  Changes in resting energy expenditure (REE) measured by indirect calorimetry
Assessment of nitrogen balance and protein breakdown in urine | -30 to 290 minutes
  Urine concentrations of urea for assessment of nitrogen balance and protein breakdown
Triglyceride responses | -30 to 290 minutes
  Plasma triglyceride
Cholesterol responses | -30 to 290 minutes
  Plasma cholesterol
Free fatty acid responses | -30 to 290 minutes
  Plasma free fatty acid

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, PhD, Principal Investigator — Center for Clinical Metabolic Research
Locations (1):
- Center for Clinical Metabolic Research, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No